CLINICAL TRIAL: NCT00446589
Title: The Effects of Ibandronate or Teriparatide Therapy on Bone Histology and Biochemical Indices in Patients on Hemodialysis With Low Bone Mineral Density
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: due to financial problems
Sponsor: Papageorgiou General Hospital (Other)
Responsible Party: Principal Investigator, Efstathios Mitsopoulos, Nephrologist, Papageorgiou General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 47b/31-1-2005
Record Dates: First submitted 2007-03-12; First posted 2007-03-13 (Estimated); Last update posted 2014-10-29 (Estimated); Status verified 2014-10

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Ibandronic Acid; Teriparatide

ARMS (2):
- F (Experimental): HD pts suffering from osteoporosis and adynamic bone disease who received teriparatide
  Interventions: Drug: teriparatide
- I (Experimental): Hemodialysis pts suffering from osteoporosis who received iv ibandronate
  Interventions: Drug: ibandronate

INTERVENTIONS:
Drug: ibandronate — iv 1mg ibandronate monthly for one year
  Arms: I
Drug: teriparatide — sc injection using a pen like device during every hemodialysis session (thrice a week)
  Arms: F

SUMMARY:
Hemodialysis patients with low bone density (total hip T-score <-2.5) will be assigned to receive teriparatide (those with histologic confirmation of adynamic bone disease) or ibandronate (subjects with increased osteoclast number on bone biopsy).

Follow-up period: one year. A second bone biopsy at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Bone mineral density (T-score<-2.5)
* Adynamic bone disease for the teriparatide group
* Increased osteoclast number on bone biopsy (high turnover) for the ibandronate group
* Calcium greater than 8.1 mg/dl

Exclusion Criteria:

* Suspected carcinoma
* Unstable clinical setting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2006-07

PRIMARY OUTCOMES:
Effects of ibandronate and teriparatide on bone mineral density and bone histology in HD patients. | one year

SECONDARY OUTCOMES:
Effects of ibandronate and teriparatide on other bone disease markers | one year

CONTACTS AND LOCATIONS:
Overall Officials: Efstathios Mitsopoulos, MD, Principal Investigator — Papageorgiou General Hospital, Thessaloniki, Greece
Locations (1):
- Papageorgiou General Hospital, Thessaloniki, Greece